CLINICAL TRIAL: NCT01463267
Title: Heart iRx This Short Non-descriptive Title is the Real Title
Brief Title: Study of Reminding to Improve Medication Adherence in Heart Failure
Acronym: Heart iRx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kent State University (Other)
Collaborators: Summa Health System (Other)
Responsible Party: Principal Investigator, Joel Hughes, Associate Professor, Kent State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 194822-4
Record Dates: First submitted 2011-09-27; First posted 2011-11-01 (Estimated); Results first posted 2020-11-27 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Heart Failure
Keywords: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Device 2 passive (Active Comparator): Device 2 will NOT remind patients to take medications
  Interventions: Behavioral: Non-reminding
- Device 2 active (Active Comparator): Device 2 will remind patients to take medications
  Interventions: Device: iPhone or pillbox
- Device 1 active (Active Comparator): Device 1 will remind patients to take their medications
  Interventions: Device: iPhone or pillbox
- Device 1 Passive (Placebo Comparator): Device 1 will NOT remind patients to take medications.
  Interventions: Behavioral: Non-reminding

INTERVENTIONS:
Device: iPhone or pillbox — People will be reminded to take their medications by a device that alerts the patient to the need to take a medication.
  Arms: Device 1 active; Device 2 active
Behavioral: Non-reminding — As a comparison, the devices will collect medication taking information without providing reminders.
  Arms: Device 1 Passive; Device 2 passive

SUMMARY:
This study is being done to look at how people manage their heart failure. The investigators are testing two medication reminder systems and the investigators want to know which one people like better. The investigators also want to see if they have any effect on ease of managing medication in individuals with heart failure.

DETAILED DESCRIPTION:
A pilot and feasibility randomized trial of two medication reminder systems for patients with heart failure (HF). The investigators believe that medication reminder systems will improve adherence and will reduce the effects of cognitive impairment on medication adherence. The investigators believe that patients will accept and use a medication reminder system, but the investigators cannot specify which system will be preferred. Each has different features which may be perceived as more or less desirable.

The investigators will enroll 60 patients with HF and randomize them to four conditions in a 2 (device 1 versus device 2) by 2 (Active versus Passive) design. After enrollment in the trial, patients will be consented and will complete pretesting at Summa Health System in the Center for Clinical Trials. They will primarily undergo brief computerized cognitive testing, complete self-report measures (e.g., quality of life, depression, self-management related social support), and will give consent for medical information to be collected from their electronic medical record. They will then be randomized to condition. In-home training will be provided regarding how to use the equipment. Medication adherence will be monitored for 28 days, followed by an in-home post-test (all pre-test measures) during which the equipment is returned.

ELIGIBILITY:
Inclusion Criteria:

* 45-90 years of age
* documented systolic or diastolic heart failure

Exclusion Criteria:

* History of neurological disorder
* moderate or severe head injury with greater than 10 min loss of consciousness
* Past or current history of severe psychiatric illness. Specifically, psychotic disorders (e.g. schizophrenia) and bipolar disorder. Potential study participants will not be excluded on the basis of managed depressive or anxiety disorder. These conditions are common in HF patients and their exclusion may limit generalizability of findings.
* 5 year past or current history of alcohol or drug abuse (defined by DSM-IV criteria)
* History of learning disorder or developmental disability (defined by DSM-IV criteria)
* Renal failure requiring dialysis
* Current home telemonitoring program to assist with HF self-management
* They do not have a land-line telephone
* Cardiac surgery < 3 months

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-11; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel W Hughes, PhD, Principal Investigator — Kent State University
Locations (1):
- Akron City Hospital, Akron, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Device 2 Passive | Device 2 Active | Device 1 Active | Device 1 Passive
Started | 15 | 15 | 15 | 15
Completed | 14 | 15 | 13 | 13
Not Completed | 1 | 0 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Device 2 Passive | Device 2 Active | Device 1 Active | Device 1 Passive | Total
Number analyzed (Participants) | 14 | 15 | 13 | 13 | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 6 | 5 | 5 | 21
  >=65 years | 9 | 9 | 8 | 8 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 69 (10.6) | 69 (10.6) | 69.6 (11.3) | 69.6 (11.3) | 69.3 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 3 | 2 | 11
  Male | 11 | 12 | 10 | 11 | 44
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14 | 15 | 13 | 13 | 55
Education [Number; unit: participants] | 14 | 15 | 13 | 13 | 55

OUTCOME MEASURES:

1. Primary Outcome: Patient Acceptance
Description: Patient ratings of their satisfaction with the device, ease of use, and other impressions. A survey was created for this study to assess individuals' evaluations of the device to which they were randomized (see Appendix 1). At the final study session, participants completed the questionnaire about their preference for the device they were assigned. The 14 items were summed into a total score reflecting their ultimate appraisal for the device. The range of possible scores was 14-70. A higher score is greater patient acceptance. Participants rated how much they agreed to each statement from strongly disagree to strongly agree. The statements assess factors such as helpfulness, improving quality of life, and satisfaction.
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Device 2 Passive | Device 2 Active | Device 1 Active | Device 1 Passive
Number analyzed (Participants) | 14 | 15 | 13 | 13
units on a scale | 33.4 (11) | 33.4 (12) | 48.7 (11) | 48.7 (12)

2. Primary Outcome: Medication Adherence
Description: The percentage of prescribed medications recorded as taken by the medication reminding device.
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: percentage of medication taken
Arm/Group | Device 2 Passive | Device 2 Active | Device 1 Active | Device 1 Passive
Number analyzed (Participants) | 14 | 15 | 13 | 13
percentage of medication taken | 76 (33) | 84 (32) | 73 (39) | 79 (33)

ADVERSE EVENTS:
Arm/Group | Device 2 Passive | Device 2 Active | Device 1 Active | Device 1 Passive
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/15 | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/14 | 0/15 | 0/13 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No